CLINICAL TRIAL: NCT06195124
Title: A Study on the Safety and Tolerability of RGL-193 Injection in Patients With Advanced Parkinson's Disease - An Open-label and Dose-escalation Clinical Trial
Brief Title: A Study on the Safety and Tolerability of RGL-193 in Patients With Advanced Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Regenelead Therapies Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chun-Feng Liu, Chief Physician, Second Affiliated Hospital of Soochow University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGL-193-IIT
Record Dates: First submitted 2023-10-14; First posted 2024-01-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Advanced Parkinson's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGL-193（low-dose）Treatment group (Experimental): Each side of the putamen received 150 μL of RGL-193, with a unilateral dose of 1.5×10^11 VG and a bilateral dose of 3.0×10^11 VG.
  Interventions: Drug: RGL-193（low-dose）
- RGL-193（high-dose）Treatment group (Experimental): Each side of the putamen received 200 μL of RGL-193, with a unilateral dose of 5.0×10^11 VG and a bilateral dose of 1.0×10^12 VG.
  Interventions: Drug: RGL-193（high-dose）

INTERVENTIONS:
Drug: RGL-193（low-dose） — Each side of the putamen received 150 μL of RGL-193, with a unilateral dose of 1.5×10^11 VG and a bilateral dose of 3.0×10^11 VG.
  Arms: RGL-193（low-dose）Treatment group
Drug: RGL-193（high-dose） — Each side of the putamen received 200 μL of RGL-193, with a unilateral dose of 5.0×10^11 VG and a bilateral dose of 1.0×10^12 VG.
  Arms: RGL-193（high-dose）Treatment group

SUMMARY:
A safety study in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation safety and tolerability study in patients with advanced Parkinson's disease

ELIGIBILITY:
Inclusion Criteria

1. The patients who voluntarily participate in the study, fully understand the content, process, and possible adverse events of the trial, can complete the study according to the requirements of the study protocol, and sign the informed consent form.
2. The patients with clinically diagnosed Parkinson's disease (as per PD diagnostic criteria, China, 2016) and the course of disease for at least 5 years at the time of screening.
3. The patient must be 45-70 years old (inclusive) on the day signing the informed consent form.
4. The patients who are receiving Levodopa treatment with clear response to Levodopa treatment.
5. The patients showing stable clinical symptoms within 1 month before baseline, with drug dosage remain the same.
6. The patients with the modified Hoehn & Yahr stage ≥ 3.
7. The patients with the score of MDS-UPDRS part III ≥ 30 in the off period.
8. There must be fluctuation of motor symptoms, which is defined as at least cumulatively 3-h off time in the awake time every day (confirmed by PD diary for 3 consecutive days).
9. The results of 18F-DOPA-PET examination shall be consistent with PD phenotype.
10. The total score of HAMD (24-item) in the screening period shall be ≤ 20 points.
11. The patients' hematological indicators and vital signs at baseline must be within the normal range, unless the values beyond the normal range have no clinical significance for whether the subjects are suitable to receive treatment with the investigational product as considered by the investigator.
12. The body weight at screening and baseline shall be 45-100 kg (inclusive), and the body mass index (BMI) shall be 18-32 kg/m2 (inclusive).
13. The subjects (including partners) shall have no fertility planning and be willing to take effective contraceptive measures during the study period (2 weeks before drug administration for female subjects) and within 6 months after administration.
14. The subjects shall have stable caregivers.

Exclusion Criteria

1. The subjects with secondary or atypical Parkinson's syndrome caused by drugs, metabolic disorders, or other reasons.
2. The subjects who have known or suspected allergies or serious adverse reactions to the ingredients of the study preparation, or those have an allergic constitution;
3. For the population with an education background of junior high school or above, the MMSE score during the screening period shall be < 23; for the population with an education background below junior high school, the MMSE score shall be < 20 during the screening period.
4. The subjects with alcoholism, acute alcohol intoxication, or drug abuse or drug dependence;
5. The subjects with a previous history of PD-related brain surgery (deep brain stimulation, thalamus destruction, etc.).
6. The subjects who have previously received any biological agents (including marketed drugs and clinical trial drugs) for PD treatment.
7. The subjects who have a history of deep venous thrombosis of lower limbs.
8. The subjects suffering from massive blood loss (more than 500 mL) due to surgery or trauma within 3 months before screening.
9. Antiplatelet and anticoagulant drugs were used within 3 months before drug administration (except aspirin (≤325mg per day));
10. The subjects with coagulation disorder, which is defined as PT > 1.2 times the upper limit of normal; a re-examination is accepted in case of a single abnormality for confirmation.
11. The subjects with obvious abnormalities in brain MRI examination, including but not limited to: more than 10 microhemorrhage foci; angiogenic edema; serious white matter demyelination (Fazekas score ≥ 3); brain contusion; encephalomalacia; aneurysm; vascular malformation, and space-occupying lesions.
12. The subjects with other major medical or nervous system diseases that may pose unacceptable risks of surgery or anesthesia, or those with any surgical contraindications.
13. The subjects unable to cooperate with the surgery or radiologic examination (DOPA PET or MRI scanning).
14. The subjects with systolic blood pressure > 160 mmHg and diastolic blood pressure > 100 mmHg in supine position in the screening period or baseline period; a re-examination is accepted in case of a single abnormality for confirmation.
15. In the screening period or baseline period, the continuous resting heart rate is < 50 bpm or > 100 bpm by repeated testing twice within 30 min.
16. The 12-lead ECG indicates remarkable abnormalities with clinical significance, including but not limited to supraventricular tachycardia, atrial fibrillation, atrial flutter, and second- or third- degree atrioventricular block, and the patients are considered not suitable to be involved in this study according to the investigator.
17. The results of ECG examination before screening or randomization indicate ECG QTcF > 450 ms. If QTcF abnormal is observed during screening, ECG examination can be repeated twice to calculate the mean QTcF value based on the 3 measurements;
18. The subjects with hepatitis B surface antigen positive, hepatitis C antibody positive (or diagnosed with active hepatitis), syphilis antibody positive, and human immunodeficiency virus (HIV) serological test positive.
19. The subjects suffering from any serious systemic infectious diseases within 1 month before screening as judged by the investigator.
20. The subjects who have received (attenuated) live vaccines within 1 month before the screening period or those who plan to receive vaccination during the trial.
21. The subjects with a history of malignant tumor within 5 years before screening, excluding the cured basal cell carcinoma of skin, papillary carcinoma of thyroid, and follicular thyroid cancer.
22. The subjects with clinically serious or unstable cardiovascular, gastrointestinal diseases, endocrine diseases, blood diseases, liver diseases, immunity diseases, metabolism diseases, urinary diseases, respiratory diseases, nervous diseases, skin diseases, mental diseases, kidney diseases, and/or other major diseases or malignant tumors that may affect the subjects' ability to participate in the study or may confuse the study results, which shall be judged by the investigator.
23. The subjects suffering from mental disorder or language disorder, resulting in inability to fully understand or cooperate, or those who are considered not appropriate for the trial according to the investigator.
24. The subjects with contraindications for magnetic resonance scanning, including but not limited to cardiac pacemakers/defibrillators and ferromagnetic metal implants (except the devices for skulls and heart approved for safe use with magnetic resonance scanners).
25. The subjects with any circumstances that may result in failures to complete the study or pose significant risks to the subjects or other factors that reduce the possibility of enrollment as considered by the investigator.
26. The subjects who have received any other investigational treatment within 3 months before screening.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the number of patients with adverse events | 26 weeks after administration
the number of patients with clinically significant change from baseline in vital signs value | 26 weeks after administration
the number of patients with clinically significant change in physical examination | 26 weeks after administration
the number of patients with clinically significant change from baseline in laboratory examination | 26 weeks after administration
the number of patients with clinically significant change from baseline in 12-ECG values | 26 weeks after administration
the number of patients with clinically significant change in brain MRI | 26 weeks after administration

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, MD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No